CLINICAL TRIAL: NCT03691974
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Effects of Fasinumab on Peripheral Nerve Function in Patients With Pain Due to Osteoarthritis of the Hip or Knee
Brief Title: Study to Evaluate the Effects of Fasinumab on Peripheral Nerve Function in Patients With Pain Due to Osteoarthritis of the Hip or Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Teva Pharmaceutical Industries, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R475-OA-1758; 2017-004921-33 (EudraCT Number)
Record Dates: First submitted 2018-09-12; First posted 2018-10-02 (Actual); Results first posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip | interventions — fasinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fasinumab (Experimental)
  Interventions: Drug: Fasinumab
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Fasinumab — Subcutaneous (SC) every four weeks (Q4W)
  Other Names: REGN475
  Arms: Fasinumab
Other: Placebo — Subcutaneous (SC) every four weeks (Q4W)
  Arms: Placebo

SUMMARY:
The primary objective of the study is to evaluate the effect of fasinumab compared to placebo on peripheral nerves in participants with pain due to Osteoarthritis (OA) of the hip or knee.

The secondary objectives of the study are to:

* Evaluate the efficacy of fasinumab compared to placebo in participants with pain due to OA of the hip or knee
* Evaluate the safety and tolerability of fasinumab compared to placebo in participants with pain due to OA of the hip or knee
* Characterize the concentrations of fasinumab in serum in participants with pain due to OA of the hip or knee
* Evaluate the immunogenicity of fasinumab in participants with pain due to OA of the hip or knee.

ELIGIBILITY:
Key Inclusion Criteria:

1. A clinical diagnosis of OA of the knee or hip based on the American College of Rheumatology criteria with radiologic evidence of OA (K-L score ≥2 for the index joint) at the screening visit
2. Moderate-to-severe pain in the index joint defined as a WOMAC average pain subscale score of ≥4 at both the screening and randomization visits
3. Willing to discontinue current pain medications and to adhere to study requirements for rescue treatments
4. A history of regular use of analgesic medications for OA pain (defined as an average of 4 days per week over the 4 weeks prior to the screening visit), including oral nonsteroidal anti-inflammatory drugs (NSAIDs), selective cyclooxygenase 2 inhibitors, opioids, paracetamol/acetaminophen, or combinations thereof
5. Consent to allow all radiographs and medical/surgical/hospitalization records of care received elsewhere prior to and during the study period to be shared with the investigator

Key Exclusion Criteria:

1. History or presence at the screening visit of non-OA inflammatory joint disease (eg, rheumatoid arthritis, lupus erythematosus, psoriatic arthritis, pseudo-gout, gout, spondyloarthropathy, polymyalgia rheumatica, joint infections within the past 5 years), Paget's disease of the spine, pelvis or femur, neuropathic disorders, multiple sclerosis, fibromyalgia, tumors or infections of the spinal cord, or renal osteodystrophy
2. History or presence on imaging of arthropathy (osteonecrosis, subchondral insufficiency fracture, rapidly progressive OA type 1 or type 2), stress fracture, recent stress fracture, neuropathic joint arthropathy, hip dislocation (prosthetic hip dislocation is eligible), knee dislocation (patella dislocation is eligible), congenital hip dysplasia with degenerative joint disease, extensive subchondral cysts, evidence of bone fragmentation or collapse, or primary metastatic tumor with the exception of chondromas or pathologic fractures during the screening period
3. Trauma to the index joint within 3 months prior to the screening visit
4. History or presence of signs or symptoms of compression neuropathy, including carpal tunnel syndrome or sciatica
5. Participant is not a candidate for Magnetic Resonance Imaging (MRI)
6. Poorly controlled diabetes
7. Known history of human immunodeficiency virus (HIV) infection
8. Known history of ocular herpes simplex virus, herpes simplex virus pneumonia, or herpes simplex virus encephalitis
9. History of poorly controlled hypertension
10. Known history of infection with hepatitis B or C virus

Note: Other protocol defined Inclusion/Exclusion apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2021-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (43):
- United States (18):
  - Regeneron Study Site, Glendale, Arizona
  - Regeneron Study Site, Phoenix, Arizona
  - Regeneron Study Site, Tucson, Arizona
  - Regeneron Study Site, Anaheim, California
  - Regeneron Study Site, Clearwater, Florida
  - Regeneron Study Site, Jacksonville, Florida
  - Regeneron Study Site, Miami, Florida
  - Regeneron Study Site, Ocoee, Florida
  - Regeneron Study Site, Orlando, Florida
  - Regeneron Study Site, Woodstock, Georgia
  - Regeneron Study Site, Chicago, Illinois
  - Regeneron Study Site, Caro, Michigan
  - Regeneron Study Site, Hartsdale, New York
  - Regeneron Study Site, Cincinnati, Ohio
  - Regeneron Study Site, Columbus, Ohio
  - Regeneron Study Site, Bellaire, Texas
  - Regeneron Study Site, Houston, Texas
  - Regeneron Study Site, San Antonio, Texas
- Poland (9):
  - Regeneron Study Site, Poznan, Greater Poland Voivodeship
  - Regeneron Study Site, Wroclaw, Lower Silesian Voivodeship
  - Regeneron Study Site, Warsaw, Masovian Voivodeship
  - Regeneron Study Site, Gdansk, Pomeranian Voivodeship
  - Regeneron Study Site, Gdynia, Pomeranian Voivodeship
  - Regeneron Study Site, Częstochowa, Silesian Voivodeship
  - Regeneron Study Site, Katowice, Silesian Voivodeship
  - Regeneron Study Site, Lodz
  - Regeneron Study Site, Lodz, Łódź Voivodeship
- United Kingdom (16):
  - Regeneron Study Site, London, Greater London
  - Regeneron Study Site, Chorley
  - Regeneron Study Site, Corby
  - Regeneron Study Site, Edgbaston
  - Regeneron Study Site, Glasgow
  - Regeneron Study Site, Hardwick
  - Regeneron Study Site, Hexham
  - Regeneron Study Site, Kenilworth
  - Regulatory Study Site, London
  - Regeneron Study Site, London
  - Regeneron Study Site, Manchester
  - Regeneron Study Site, Northwood
  - Regeneron Study Site, Peterborough
  - Regeneron Study Site, Reading
  - Regeneron Study Site, Shipley
  - Regeneron Study Site, Waterloo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1604 participants were screened, out of which 180 were randomized into the study from 47 centers in North America and Europe.
Pre-assignment Details: Participants who met the eligibility criteria were randomized in 1:1 ratio to receive Fasinumab or matched placebo.
Groups:
- Fasinumab-matching Placebo: Participants received Fasinumab-matching placebo subcutaneously (SC) every 4 weeks (Q4W) from Day 1 through Week 12 of the 16-week treatment period.
- Fasinumab 1 mg SC Q4W: Participants received Fasinumab 1 milligram (mg) SC Q4W from Day 1 through Week 12 of the 16-week treatment period.
Period: Overall Study
Arm/Group | Fasinumab-matching Placebo | Fasinumab 1 mg SC Q4W
Started | 89 | 91
Completed | 67 | 75
Not Completed | 22 | 16
Not completed — Physician Decision | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 11 | 9
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 8 | 7

BASELINE CHARACTERISTICS:
Groups:
- Fasinumab-matching Placebo: Participants received Fasinumab-matching placebo SC Q4W from Day 1 through Week 12 of the 16-week treatment period.
- Fasinumab 1 mg SC Q4W: Participants received Fasinumab 1 mg SC Q4W from Day 1 through Week 12 of the 16-week treatment period.
- Total: Total of all reporting groups
Arm/Group | Fasinumab-matching Placebo | Fasinumab 1 mg SC Q4W | Total
Number analyzed (Participants) | 89 | 91 | 180
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.4 (7.9) | 62.9 (9.1) | 62.7 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 59 | 122
  Male | 26 | 32 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 8 | 13
  Not Hispanic or Latino | 83 | 81 | 164
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 8 | 13
  White | 80 | 78 | 158
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Peroneal Motor Nerve Conduction Velocity [Mean (Standard Deviation); unit: Meters per Second (m/sec)] — Peroneal motor nerve conduction velocity was evaluated by electrical stimulation of the nerve and recorded the compound muscle action potential from surface electrodes overlying a muscle supplied by the nerve. Population: The safety analysis set (SAF) included all randomized participants who received any study drug and was based on the treatment received (as treated).
  Meters per Second (m/sec)
    number analyzed (Participants) | 88 | 91 | 179
    (all) | 46.86 (4.17) | 46.80 (3.88) | 46.83 (4.02)
Peroneal Motor Nerve Action Potential Amplitude - Ankle [Mean (Standard Deviation); unit: Millivolts (mV)] — Peroneal motor nerve action potential amplitude was evaluated at ankle by electrical stimulation of the nerve and recorded the compound muscle action potential from surface electrodes overlying a muscle supplied by the nerve. Population: The SAF included all randomized participants who received any study drug and was based on the treatment received (as treated).
  Millivolts (mV)
    number analyzed (Participants) | 88 | 91 | 179
    (all) | 4.75 (2.01) | 4.67 (1.70) | 4.71 (1.85)
Sural Sensory Nerve Conduction Velocity [Mean (Standard Deviation); unit: m/sec] — Sural sensory nerve conduction velocity was evaluated by electrically stimulating sensory fibers and recorded the nerve action potential at a point further along that nerve. Population: The SAF included all randomized participants who received any study drug and was based on the treatment received (as treated).
  m/sec
    number analyzed (Participants) | 88 | 91 | 179
    (all) | 52.35 (8.52) | 52.49 (8.28) | 52.42 (8.37)
Sural Sensory Nerve Action Potential Amplitude [Mean (Standard Deviation); unit: Microvolts (mcV)] — Sural sensory nerve action potential amplitude was evaluated by electrically stimulating sensory fibers and recorded the nerve action potential at a point further along that nerve. Population: The SAF included all randomized participants who received any study drug and was based on the treatment received (as treated).
  Microvolts (mcV)
    number analyzed (Participants) | 88 | 91 | 179
    (all) | 9.67 (4.79) | 9.95 (5.67) | 9.82 (5.24)
Ulnar Sensory Nerve Conduction Velocity [Mean (Standard Deviation); unit: m/sec] — Ulnar sensory nerve conduction velocity was evaluated by electrically stimulating sensory fibers and recorded the nerve action potential at a point further along that nerve. Population: The SAF included all randomized participants who received any study drug and was based on the treatment received (as treated).
  m/sec
    number analyzed (Participants) | 88 | 91 | 179
    (all) | 56.03 (6.58) | 56.24 (7.45) | 56.14 (7.02)
Ulnar Sensory Nerve Action Potential Amplitude [Mean (Standard Deviation); unit: mcV] — Ulnar sensory nerve action potential amplitude was evaluated by electrically stimulating sensory fibers and recorded the nerve action potential at a point further along that nerve. Population: The SAF included all randomized participants who received any study drug and was based on the treatment received (as treated).
  mcV
    number analyzed (Participants) | 88 | 91 | 179
    (all) | 19.18 (9.68) | 18.47 (10.20) | 18.82 (9.92)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Peroneal Motor Nerve Conduction Velocity at Week 16
Description: Peroneal motor nerve conduction velocity was evaluated by electrical stimulation of the nerve and recorded the compound muscle action potential from surface electrodes overlying a muscle supplied by the nerve. Change from baseline in peroneal motor nerve conduction velocity at Week 16 was reported.
Time Frame: Baseline, Week 16
Population: The SAF included all randomized participants who received any study drug and was based on the treatment received (as treated). Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: m/sec
Arm/Group | Fasinumab-matching Placebo | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 69 | 84
m/sec | -0.2 (0.46) | 0.2 (0.42)
Statistical Analysis 1: Comparison: Fasinumab-matching Placebo vs Fasinumab 1 mg SC Q4W; Test type: Superiority; p = 0.4192, Mixed Model for Repeated Measures (MMRM) — Analyses are based on Mixed Model for Repeated Measures (MMRM) model with terms for baseline nerve conduction test score, treatment, screening Kellgren-Lawrence score, index joint, visit, and treatment by visit interaction; Least Square (LS) Mean Difference = 0.4, 95% CI 2-sided [-0.55 to 1.32]

2. Primary Outcome: Change From Baseline in Peroneal Motor Nerve Action Potential Amplitude at Week 16
Description: Peroneal motor nerve action potential amplitude was evaluated at ankle by electrical stimulation of the nerve and recorded the compound muscle action potential from surface electrodes overlying a muscle supplied by the nerve. Change from baseline in peroneal motor nerve action potential amplitude at Week 16 was reported.
Time Frame: Baseline, Week 16
Population: SAF included all randomized participants who received any study drug and was based on the treatment received (as treated). Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: mV
Arm/Group | Fasinumab-matching Placebo | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 69 | 84
mV | -0.2 (0.20) | 0.2 (0.19)
Statistical Analysis 1: Comparison: Fasinumab-matching Placebo vs Fasinumab 1 mg SC Q4W; Test type: Superiority; p = 0.0521, MMRM — Analyses are based on MMRM model with terms for baseline nerve conduction test score, treatment, screening Kellgren-Lawrence score, index joint, visit, and treatment by visit interaction; LS Mean Difference = 0.4, 95% CI 2-sided [-0.00 to 0.80]

3. Primary Outcome: Change From Baseline in Sural Sensory Nerve Conduction Velocity at Week 16
Description: Sural sensory nerve conduction velocity was evaluated by electrically stimulating sensory fibers and recorded the nerve action potential at a point further along that nerve. Change from baseline in sural sensory nerve conduction velocity at Week 16 was reported.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: m/sec
Arm/Group | Fasinumab-matching Placebo | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 69 | 84
m/sec | -2.9 (0.90) | -1.6 (0.83)
Statistical Analysis 1: Comparison: Fasinumab-matching Placebo vs Fasinumab 1 mg SC Q4W; Test type: Superiority; p = 0.1593, MMRM — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 1.3, 95% CI 2-sided [-0.52 to 3.15]

4. Primary Outcome: Change From Baseline in Sural Sensory Nerve Action Potential Amplitude at Week 16
Description: Sural sensory nerve action potential amplitude was evaluated by electrically stimulating sensory fibers and recorded the nerve action potential at a point further along that nerve. Change from baseline in sural sensory nerve action potential amplitude at Week 16 was reported.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mcV
Arm/Group | Fasinumab-matching Placebo | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 69 | 84
mcV | 0.5 (0.69) | 0.3 (0.64)
Statistical Analysis 1: Comparison: Fasinumab-matching Placebo vs Fasinumab 1 mg SC Q4W; Test type: Superiority; p = 0.7757, MMRM — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.2, 95% CI 2-sided [-1.59 to 1.19]

5. Primary Outcome: Change From Baseline in Ulnar Sensory Nerve Conduction Velocity at Week 16
Description: Ulnar sensory nerve conduction velocity was evaluated by electrically stimulating sensory fibers and recorded the nerve action potential at a point further along that nerve. Change from baseline in ulnar sensory nerve conduction velocity at Week 16 was reported.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: m/sec
Arm/Group | Fasinumab-matching Placebo | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 69 | 84
m/sec | -0.7 (0.74) | -1.1 (0.68)
Statistical Analysis 1: Comparison: Fasinumab-matching Placebo vs Fasinumab 1 mg SC Q4W; Test type: Superiority; p = 0.6063, MMRM — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.4, 95% CI 2-sided [-1.87 to 1.09]

6. Primary Outcome: Change From Baseline in Ulnar Sensory Nerve Action Potential Amplitude at Week 16
Description: Ulnar sensory nerve action potential amplitude was evaluated by electrically stimulating sensory fibers and recorded the nerve action potential at a point further along that nerve. Change from baseline ulnar sensory nerve action potential amplitude at Week 16 was reported.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mcV
Arm/Group | Fasinumab-matching Placebo | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 69 | 84
mcV | 2.4 (1.21) | 1.4 (1.12)
Statistical Analysis 1: Comparison: Fasinumab-matching Placebo vs Fasinumab 1 mg SC Q4W; Test type: Superiority; p = 0.4203, MMRM — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -1.0, 95% CI 2-sided [-3.30 to 1.39]

7. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score at Week 16
Description: WOMAC pain subscale was a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis in the index joint (knee or hip) in past 48 hours. It was calculated as the mean of the scores from the 5 individual questions scored on a numerical rating scale (NRS) of 0 (no pain) to 10 (higher pain), where higher scores indicated higher pain. Total score range for WOMAC pain subscale score is 0 to 10, where higher scores indicate higher pain. A negative change from baseline indicated improvement. Change from baseline in WOMAC Pain subscale score at Week 16 was reported.
Time Frame: Baseline, Week 16
Population: FAS included all randomized participants and was based on the treatment allocated (as randomized). Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Fasinumab-matching Placebo | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 54 | 67
Score on a Scale | -1.19 (0.359) | -2.52 (0.335)
Statistical Analysis 1: Comparison: Fasinumab-matching Placebo vs Fasinumab 1 mg SC Q4W; Test type: Superiority; p = 0.0010, MMRM — Analyses are based on multiple imputation with MMRM model with terms for baseline WOMAC subscale score, treatment, screening Kellgren-Lawrence score, index joint, visit, and treatment by visit interaction; LS Mean Difference = -1.33, 95% CI 2-sided [-2.123 to -0.538]

8. Secondary Outcome: Change From Baseline in WOMAC Physical Function Subscale Score at Week 16
Description: Physical function referred to subject's ability to move around and perform usual activities of daily living. The WOMAC physical function subscale was a 17-item questionnaire used to assess the degree of difficulty experienced due to osteoarthritis in index joint (knee or hip) during past 48 hours. It was calculated as mean of the scores from 17 individual questions scored on a NRS of 0 (no difficulty) to 10 (extreme difficulty), where higher scores indicated worse function. Total score range for WOMAC physical function subscale score is 0 (no difficulty) to 10 (extreme difficulty), where higher scores indicate worse function. A negative change from baseline indicated improvement. Change from baseline in WOMAC physical function subscale score at Week 16 was reported.
Time Frame: Baseline, Week 16
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Fasinumab-matching Placebo | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 54 | 66
Score on a Scale | -0.83 (0.366) | -2.24 (0.341)
Statistical Analysis 1: Comparison: Fasinumab-matching Placebo vs Fasinumab 1 mg SC Q4W; Test type: Superiority; p = 0.0005, MMRM — Analyses were based on multiple imputation with MMRM model with terms for baseline WOMAC subscale score, treatment, screening Kellgren-Lawrence score, index joint, visit, and treatment by visit interaction; LS Mean Difference = -1.42, 95% CI 2-sided [-2.212 to -0.625]

9. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant administered a study drug which may or may not have a causal relationship with the study drug. A serious adverse event (SAE) was defined as any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. TEAE was defined as an AE with an onset that occurs after receiving study drug. Any TEAE included participants with both serious and non-serious TEAEs. Number of participants with TEAEs were reported.
Time Frame: Baseline up to Week 16
Population: SAF included all randomized participants who received any study drug and was based on the actual treatment received (as treated).
Measure: Count of Participants; unit: Participants
Arm/Group | Fasinumab-matching Placebo | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 88 | 91
Participants | 57 | 63

10. Secondary Outcome: Number of Adjudicated Arthropathy (AA) Events
Description: AA was a composite term that encompasses the following conditions: Rapidly progressive Osteoarthritis (OA) type 1 and 2, Subchondral insufficiency fractures, and Primary Osteonecrosis confirmed by an arthropathy adjudication committee. Number of confirmed AA events from baseline up to follow-up (Week 36) were reported.
Time Frame: Baseline up to follow-up (Week 36)
Population: as for outcome 9
Measure: Number; unit: Adjudicated Arthropathy (AA) Events
Arm/Group | Fasinumab-matching Placebo | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 88 | 91
Adjudicated Arthropathy (AA) Events | 0 | 4

11. Secondary Outcome: Number of AA Events Meeting Destructive Arthropathy (DA) Criteria
Description: AAs were evaluated to determine if they met Destructive Arthropathy (DA) criteria. DA is a unique clinical form of rapidly destructive arthropathy over and above that seen in the normal progression of OA. DA criteria can be associated with Rapidly Progressive OA type 2, Subchondral Insufficiency fracture, and Primary Osteonecrosis confirmed by an arthropathy adjudication committee. Number of confirmed AA events meeting DA criteria from baseline up to follow-up (Week 36) were reported.
Time Frame: Baseline up to follow-up (Week 36)
Population: SAF included all randomized participants who received any study drug and was based on the actual treatment received (as treated). "Overall Number of Participants Analyzed" signifies those participants who had confirmed AA events.
Measure: Number; unit: Destructive Arthropathy (DA) Events
Arm/Group | Fasinumab-matching Placebo | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 0 | 4
Destructive Arthropathy (DA) Events |  | 0

12. Secondary Outcome: Number of Sympathetic Nervous System (SNS) Dysfunction Events
Description: Potential events of SNS dysfunction were monitored throughout the study through physical examination, AE reporting, assessment of orthostatic hypotension, and the Survey of Autonomic Symptoms. Sympathetic nervous system dysfunction was diagnosed after consultation with an appropriate specialist, such as a neurologist and/or cardiologist. Number of SNS dysfunction events from baseline up to follow-up (Week 36) were reported.
Time Frame: Baseline up to follow-up (Week 36)
Population: as for outcome 9
Measure: Number; unit: SNS Dysfunction Events
Arm/Group | Fasinumab-matching Placebo | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 88 | 91
SNS Dysfunction Events | 0 | 0

13. Secondary Outcome: Number of Peripheral Sensory Adverse Events (AEs) That Require a Neurology Consultation
Description: Any peripheral sensory AE (for example [e.g.], paraesthesia and hypoaesthesia) that required a neurology consultation. Number of peripheral sensory adverse events from baseline up to follow-up (Week 36) were reported.
Time Frame: Baseline up to follow-up (Week 36)
Population: as for outcome 9
Measure: Number; unit: Peripheral Sensory Adverse Events (AEs)
Arm/Group | Fasinumab-matching Placebo | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 88 | 91
Peripheral Sensory Adverse Events (AEs)
  Carpal tunnel syndrome | 4 | 4
  Decreased vibratory sense | 0 | 3
  Hypoaesthesia | 1 | 0
  Neuropathy peripheral | 1 | 3
  Paraesthesia | 1 | 2

14. Secondary Outcome: Number of All-Cause Joint Replacement (JR) Surgery Events
Description: All joint replacement surgery events regardless of cause.
Time Frame: Baseline up to follow-up (Week 36)
Population: as for outcome 9
Measure: Number; unit: Joint Replacement (JR) Surgery Events
Arm/Group | Fasinumab-matching Placebo | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 88 | 91
Joint Replacement (JR) Surgery Events | 4 | 5

15. Secondary Outcome: Number of Joint Replacement (JR) Surgery Events Reported at Telephone Survey After Last Dose of Study Drug
Description: An end of study phone contact was conducted approximately 52 weeks following the last dose of study drug (Week 64) to evaluate the number of participants who had undergone or were scheduled for JR surgery.
Time Frame: Baseline up to EOS (Week 64)
Population: as for outcome 9
Measure: Number; unit: Joint Replacement (JR) Surgery Events
Groups:
- Placebo: Participants received SC injection of placebo matched to Fasinumab Q4W on Day 1, Weeks 4, 8 and 12.
- Fasinumab 1 mg SC Q4W: Subjects received SC injection of Fasinumab at a dose of 1 mg Q4W on Day 1, Weeks 4, 8 and 12.
Arm/Group | Placebo | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 88 | 91
Joint Replacement (JR) Surgery Events | 1 | 0

16. Secondary Outcome: Serum Concentration of Functional Fasinumab
Description: Serum concentrations of functional Fasinumab were reported.
Time Frame: Baseline, Week 1, 2, 4, 8, 12, 16 and 36
Population: The Pharmacokinetic (PK) Analysis Set included all treated participants who received any study drug and who had at least 1 non-missing drug concentration result following the first dose of study drug. Here, "Number Analyzed" signifies those participants who were evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: Milligrams per Liter (mg/L)
Arm/Group | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 91
Milligrams per Liter (mg/L)
  Baseline | 0 (0)
  Week 1: number analyzed (Participants) | 84
  Week 1 | 0.0864 (0.029)
  Week 2: number analyzed (Participants) | 87
  Week 2 | 0.0820 (0.025)
  Week 4: number analyzed (Participants) | 85
  Week 4 | 0.0525 (0.018)
  Week 8: number analyzed (Participants) | 84
  Week 8 | 0.0780 (0.0326)
  Week 12: number analyzed (Participants) | 81
  Week 12 | 0.0802 (0.040)
  Week 16: number analyzed (Participants) | 76
  Week 16 | 0.0824 (0.049)
  Week 36: number analyzed (Participants) | 11
  Week 36 | 0 (0)

17. Secondary Outcome: Number of Participants With At-least One Positive Anti-Drug Antibody (ADA)
Description: Samples for ADA evaluation were collected at baseline and at subsequent study visits. ADA variables included ADA status (+/-) and titer as follows: Total participants negative in ADA assay at all time points analyzed. Pre-existing immunoreactivity- positive response at baseline with all post-dose results negative/positive response at baseline with all post-dose responses less than 9-fold over baseline titer levels. Treatment emergent - post-dose positive result when baseline results were negative. Persistent - A positive result detected in at least/ more 2 consecutive post baseline samples separated by at least a 16-week post baseline period, with no negative results in-between. Indeterminate - A positive result at the last collection time point analyzed only. Transient - Not persistent or indeterminate regardless of any missing samples. Treatment boosted- positive response in ADA assay post first dose that is greater than/equal 9-fold over baseline level when baseline is positive.
Time Frame: Baseline up to follow-up period (Week 36)
Population: The anti-drug antibody (ADA) analysis set included all treated participants who received any study drug and had at least 1 qualified (non-missing) ADA result following the first dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Fasinumab-matching Placebo | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 80 | 87
Participants
  Pre-Existing Immunoreactivity | 1 | 0
  Treatment-Boosted Response | 0 | 0
  Treatment-Emergent Response | 0 | 0
  Treatment-Emergent: Persistent | 0 | 0
  Treatment-Emergent: Transient | 0 | 0
  Treatment-Emergent: Indeterminate | 0 | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to 24 weeks post the last dose of study drug (up to Week 36)
Description: Reported adverse events (AEs) are AEs that developed/worsened from the time of the first administration of study drug until the end of the follow up period (Week 36).
Arm/Group | Fasinumab-matching Placebo | Fasinumab 1 mg SC Q4W
All-Cause Mortality (participants affected / at risk) | 0/88 | 0/91
Serious Adverse Events (participants affected / at risk) | 6/88 | 3/91
Other Adverse Events (participants affected / at risk) | 49/88 | 55/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fasinumab-matching Placebo (N=88) | Fasinumab 1 mg SC Q4W (N=91)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Rapidly progressive osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lung squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fasinumab-matching Placebo (N=88) | Fasinumab 1 mg SC Q4W (N=91)
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 (27) | 24 (44)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0)
Headache (Nervous system disorders) | 15 (26) | 13 (22)
Nerve conduction studies abnormal (Investigations) | 17 (17) | 10 (13)
Nasopharyngitis (Infections and infestations) | 6 (8) | 8 (10)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 5 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (8) | 6 (7)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (6)
Dizziness (Nervous system disorders) | 3 (3) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 5 (6) | 5 (5)
Urinary tract infection (Infections and infestations) | 4 (5) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights

DOCUMENTS (2):
  • Study Protocol (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/74/NCT03691974/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/74/NCT03691974/SAP_001.pdf